CLINICAL TRIAL: NCT03988153
Title: Efficacy of Probiotic Milk Formula on Blood Lipid and Intestinal Function in Mild Hypercholesterolemic Volunteers: A Placebo-control, Randomized Clinical Trial
Brief Title: Efficacy of Probiotic Milk Formula on Blood Lipid and Intestinal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Chin Kun Wang, Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS08006
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Healthy
Keywords: Probiotics; cholesterol; LDL-c; Hypercholesterolemic; Fecal movement

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, randomized parallel clinical trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Milk Formula (PMF) (Experimental): Twenty subjects should drink 200 mL of PMF (30 gm mixed with 200 mL of water) before breakfast and dinner (2 times/day) for 10 weeks
  Interventions: Combination Product: Probiotic Milk Formula
- Skimmed Milk Formula (Placebo Comparator): Twenty subjects should drink 200 mL of skimmed milk drink (30 gm mixed with 200 mL of water) before breakfast and dinner (2 times/day) for 10 weeks
  Interventions: Combination Product: Probiotic Milk Formula

INTERVENTIONS:
Combination Product: Probiotic Milk Formula — Drink 200 mL of PMF for 10 weeks and followed by 2 weeks of follow up period for monitor any adverse effect

SUMMARY:
Probiotic contained milk formula (PMF) intervention for 10 weeks considerably improves gastrointestinal function by modulating fecal movement, intestinal microflora as well as decrease cholesterol and thus help in the management of hypercholesterolemia.

DETAILED DESCRIPTION:
Current randomized placebo-controlled, double-blind was designed to assess the effect of probiotic contained milk formula (PMF) on lipid profile and intestinal function in healthy mild hypercholesterolemic subjects. Totally forty healthy mild hypercholesterolemic subjects (180-220 mg/dL) were randomly chosen and divided into two groups as placebo or experimental group. All the subjects were requested to drink either PMF (experimental) or skimmed milk drink formula-Placebo (30 gm mixed with 200 mL of water) for 10 weeks and continued by 2 weeks of the follow-up period. Supplementation of PMF for 10 weeks significantly improved (p< 0.05) the fecal weight, fecal movement (decreased fecal GI passing time) by improving intestinal microflora (increasing beneficial bacterial species like Lactobacillus, Bifidobacterium spp) and Lag time of LDL oxidation. In addition, intake of PMF substantially reduced (p< 0.05) the levels of total cholesterol (TC) and low-density lipoprotein cholesterol (LDL-c) and thus showcasing its cardioprotective efficacy. Therefore PMF is recommended for the management of hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* healthy mild hypercholesterolemic subjects (180-220 mg/dL)

Exclusion Criteria:

* Subjects who took antibiotics or supplements (vitamins or minerals), probiotics (especially dairy products), Subjects suffering from severe gastrointestinal, cardiovascular, hepatic or renal disorders, Lactating or pregnant women, chain smokers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-11-10 (Actual); Primary Completion 2011-03-15 (Actual); Study Completion 2011-04-20 (Actual)

PRIMARY OUTCOMES:
Fecal Characteristics | 12 weeks
  Intervention with PMF to check the change in fecal weight (mg)
Intestinal microflora | 12 weeks
  Intervention with PMF to check the change in fecal Lactobacillus spp content (1 mg)

SECONDARY OUTCOMES:
Lipid profile | 12 weeks
  Intervention with PMF to check the changes in total cholesterol (mg/dl)
Lag time of LDL oxidation | 12 weeks (5 min incubation)
  Intervention with PMF to check the LDL oxidation time (minutes)

IPD SHARING:
Plan to Share IPD: No